CLINICAL TRIAL: NCT05354921
Title: Hip Fracture Patient and the Use of IndwElling vs IntermittEnt Catheterization Pilot Study
Brief Title: Indwelling vs Intermittent Catheterization Pilot Study
Acronym: PEE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20220067-01H
Record Dates: First submitted 2022-04-11; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Urogenital; Urinary Tract Infections; Hip Fractures; Catheter Complications
MeSH Terms: conditions — Urinary Tract Infections; Hip Fractures | interventions — Catheters, Indwelling; Intermittent Urethral Catheterization

STUDY DESIGN:
Masking Description: A clinical research coordinator that is blinded to the arm patients are randomized to will be responsible for recording all outcome measures of interest prospectively in the study's database from the patient's electronic medical records.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indwelling (Experimental): Foley catheterization upon admission and removed the morning following surgery.
  Interventions: Device: Indwelling Catheter
- Intermittent (Experimental): Intermittent catheterization when post-void residual volume is greater than 400 mL.
  Interventions: Device: Intermittent Catheterization

INTERVENTIONS:
Device: Indwelling Catheter — Patients in the experimental group will receive foley catheter upon admission, aseptically. The catheter will be discontinued on the morning following surgery. At TOH most (>75%) hip fractures are treated within 48 hours of admission and 95% within 72 hours and hence the indwelling catheter is likely to stay in place for 3-4 days.
  Arms: Indwelling
Device: Intermittent Catheterization — Patients randomized to the intermittent catheterization group will have their PVR monitored every 8 hours pre-operatively. If PVR>400 mL, an intermittent catheter will be used. If PVR> 400 mL greater than 3 times pre-operatively, an indwelling catheter will be placed the fourth time. The indwelling catheter will be removed the morning of post-op day 1.
  It is expected that a small percentage of patients in either group will not have a PVR>400 mL preoperatively.
  These patients will not be catheterized but will remain in the study. Post-operatively, both treatment groups will have their PVR monitored for 24 hours, or until PVR is less than 200 mL. If PVR>400 mL and the patient is not able to void further, intermittent catheterization will be done every six hours as needed. If post-operative PVR>400 mL greater than 3 times post-operatively, an indwelling catheter will be placed the fourth time.
  Arms: Intermittent

SUMMARY:
The primary aim of the proposed pilot feasibility is to determine whether it is feasible to recruit patients with a hip fracture into a prospective study and randomize them to either indwelling or intermittent catheterization. The study hypothesis is that the investigators would be able to show that this study can be incorporated into clinical practice, with satisfactory rate of patient recruitment and retention. Thus, the investigators would be able to compete this pilot study trial and proceed towards a multi-center trial.

DETAILED DESCRIPTION:
The primary aim of the proposed pilot feasibility is to determine whether it is feasible to recruit patients with a hip fracture into a prospective study and randomize them to either indwelling or intermittent catheterization.

The study hypothesis is that the investigators would be able to show that this study can be incorporated into clinical practice, with satisfactory rate of patient recruitment and retention. Thus, the investigators would be able to compete this vanguard trial and proceed towards a multi-center trial.

Secondary objectives would be related to safety and patient activity that would be important endpoints for the definitive, large scale trial. These would include the following:

1. Is short term indwelling catheter use associated with reduced incidence of UTI compared to clean intermittent catheterization in patients with hip fracture.
2. How does patient experience compare between these two forms of treatment?

Eligible patients will be approached for consent at admission and, if willing to participate, will be randomized into Group A or Group B using a web-based, computer-generated randomization with permuted blocks of varying sizes.

Data Collection will include:

* Urinary symptoms at admission, pre-fracture
* Date and time of catheter insertion (indwelling or not)
* Date and time of surgery
* Type of anesthesia used
* Date and time of catheter removal
* Number of catheterizations performed during hospital stay
* Type of Antibiotic cover during per-operative period (typically 3 doses provided perioperatively)

A clinical research coordinator (CRC) will oversee study recruitment and assess number of study participants to the total number of patients admitted with a hip fracture which will allow for documentation of ability to recruit into the study. Furthermore, the CRC will prospectively record each patent's journey to assess whether enrolled patients are receiving the treatment they are randomized to. All enrolled patients will be asked to fill in a patient satisfaction score that has been in use already at our institution.

A CRC, blinded to the arm patients were randomized to, will be responsible for recording all outcome measures of interest prospectively in the study's database from the participant's electronic medical records. Validity of data extraction will be tested for a randomly selected 10% of the cohort by a second evaluator (CRC not previously involved in the study).

Data analyses will include:

Descriptive Statistics: Given the feasibility purpose of the vanguard trial, descriptive statistics will be used to summarize demographics and baseline prognostic factors of participants allocated to the two trial arms.

Analysis of Primary Outcome: Our primary endpoint is the rate of enrolment to ensure the ability to undertake a larger multi-centered trial. An average rate of 10 patients/month or greater will be considered as ideal for establishing feasibility. An enrollment of less than 5 patients/month will likely jeopardize the ability to feasibly recruit for the larger trial. Whereas, average monthly enrolment of 5 to 10 patients will require a re-evaluation of our recruitment strategy, intervention specifications, and/or eligibility criteria to improve enrolment.

Analysis of Secondary Outcomes: Given the vanguard nature of this trial, the investigators will not undertake inferential analyses of our secondary outcomes but rather these patients will be carried forward into the larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture (intertrochanteric, femoral neck, femoral head, sub-trochanteric) confirmed by imaging
* Age ≥50 years
* Operative treatment planned
* Admitted under Orthopaedic Surgery
* Willing and able to sign consent (substitute decision maker)

Exclusion Criteria:

* Periprosthetic hip fracture
* Polytrauma
* Multiple fractures of the lower limbs
* Previous lower urinary tract surgery
* Known (past or current) urogenital cancer (prostate, bladder)
* Urinary tract infection prior to randomization
* Indwelling catheter present on admission (chronic or placed at previous acute setting)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility - Enrollment | One year
  Number of participants enrolled and willingness of participants to be randomized Comparing the Number of patients screened compared to the number of patients meeting eligibility criteria.
  Tracking crossover between the treatment groups, participant retention, and follow-up rates.
Study Feasibility - Screening | One year
  Number of patients screened and number meeting eligibility
Study Feasibility - Retention | One year
  Participant retention rate in study
Study Feasibility - Follow-up | One year
  Rates of participant follow-up

SECONDARY OUTCOMES:
Safety-Related Outcomes - Rates of UTI | 30 days
  Number of patients who present with a post-operative UTI within 30 days of catheterization
Safety-Related Outcomes - Rates of POUR | 30 days
  Number of patients who present with post-operative POUR within 30 days of catheterization
patient experience questionnaire | pre-operatively, and post-operative day six or at discharge
  the patient experience questionnaire, created by the principal investigator of the study, will be used to assess patients level of urogenital pain and discomfort and satisfaction with catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: George Grammatopoulos, MD, Principal Investigator — The Ottawa Hospital; Steven Papp, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Health Quality Ontario, M.o.H.a.L.-T.C., Quality Based Procedures Clinical Handbook for Hip Fracture. 2013.
- [Result] Dodd AC, Bulka C, Jahangir A, Mir HR, Obremskey WT, Sethi MK. Predictors of 30-day mortality following hip/pelvis fractures. Orthop Traumatol Surg Res. 2016 Oct;102(6):707-10. doi: 10.1016/j.otsr.2016.05.016. Epub 2016 Aug 3. PMID 27496661
- [Result] Skelly JM, Guyatt GH, Kalbfleisch R, Singer J, Winter L. Management of urinary retention after surgical repair of hip fracture. CMAJ. 1992 Apr 1;146(7):1185-9. PMID 1555145
- [Result] Smith NK, Albazzaz MK. A prospective study of urinary retention and risk of death after proximal femoral fracture. Age Ageing. 1996 Mar;25(2):150-4. doi: 10.1093/ageing/25.2.150. PMID 8670545
- [Result] Hedstrom M, Grondal L, Ahl T. Urinary tract infection in patients with hip fractures. Injury. 1999 Jun;30(5):341-3. doi: 10.1016/s0020-1383(99)00094-7. PMID 10505128
- [Result] Kamdar A, Yahya A, Thangaraj L. Retrospective observational study of the incidence of short-term indwelling urinary catheters in elderly patients with neck of femur fractures. Geriatr Gerontol Int. 2009 Jun;9(2):131-4. doi: 10.1111/j.1447-0594.2008.00490.x. PMID 19740355
- [Result] Schneider MA. Prevention of catheter-associated urinary tract infections in patients with hip fractures through education of nurses to specific catheter protocols. Orthop Nurs. 2012 Jan-Feb;31(1):12-8. doi: 10.1097/NOR.0b013e3182419619. PMID 22278644
- [Result] Gould CV, Umscheid CA, Agarwal RK, Kuntz G, Pegues DA; Healthcare Infection Control Practices Advisory Committee. Guideline for prevention of catheter-associated urinary tract infections 2009. Infect Control Hosp Epidemiol. 2010 Apr;31(4):319-26. doi: 10.1086/651091. No abstract available. PMID 20156062
- [Result] Thomas S, Harris N, Dobransky J, Grammatopoulos G, Gartke K, Liew A, Papp S. Urinary catheter use in patients with hip fracture: Are current guidelines appropriate? A retrospective review. Can J Surg. 2021 Nov 25;64(6):E630-E635. doi: 10.1503/cjs.014620. Print 2021 Nov-Dec. PMID 34824151
- [Result] Excellence, N.I.f.H.a.C., Hip fracture: management. 2011.